CLINICAL TRIAL: NCT00111891
Title: A Dose Ranging Study to Evaluate the Tolerability of MK0524 (Niacin (+) Laropiprant) and Its Effects on Niacin-Induced Acute Flushing in Lipid Clinic Patients and/or Normal Healthy Subjects
Brief Title: An Investigational Drug Study Evaluating a Novel Approach to Treat Dyslipidemia (0524A-032)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524-032; MK0524A-032; 2005_032
Record Dates: First submitted 2005-05-26; First posted 2005-05-27 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: niacin (+) laropiprant
  Other Names: MK0524A
Drug: Comparator: placebo (unspecified)

SUMMARY:
This is a 3-week trial in normal healthy or lipid clinic patients studying a novel approach to treating dyslipidemia.

DETAILED DESCRIPTION:
The duration of treatment is 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (ages 25-75)

Exclusion Criteria:

* A condition which, in the opinion of the investigator, might pose a risk to the patient or interfere with participating in the study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2005-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Acute cutaneous symptoms induced by niacin for 7 days. | 7 days

SECONDARY OUTCOMES:
Tolerability | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html